CLINICAL TRIAL: NCT03746145
Title: A Counter Measure for the Effects of Immune and Microbiome Changes in Environments With Limited ANtigen Diversity (ICELAND-TWO) - a Randomized Double Blind Controlled Pilot Study With Bifidobacterium Longum 1714
Brief Title: A Counter Measure for the Effects of Immune and Microbiome Changes in Environments With Limited ANtigen Diversity (ICELAND-TWO)
Acronym: ICELAND-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Dr. Isabelle Mack, Co-PI, University Hospital Tübigen (Unknown); Dr. Claude Lambert, University Hospital of Saint-Etienne (Unknown); Dr. John Penders, Maastricht University Medical Center (Unknown); Dr. Joël Doré, Institut National de la Recherche Agronomique (Unknown); European Space Agency (Other)
Responsible Party: Principal Investigator, Prof. Dr. Paul Enck, Director of Research, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ICELAND-2
Record Dates: First submitted 2018-11-08; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Confinement and Isolation
Keywords: probiotics; microbiota; gastrointestinal; immune system; immunology; stress; Bifidobacterium; hypoxia; confinement; isolation
MeSH Terms: conditions — Hypoxia | interventions — stearic acid

STUDY DESIGN:
Intervention Model Description: During the entire winter over (WO) period, from arrival at COCORDIA until departure (1 year), participants receive 2g nutritional supplement powder (sachet, containing 10e11 CFU Bifidobacterium longum 1714 or placebo) once every day, to be taken in the morning with breakfast throughout the year.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium longum 1714 (Experimental): Participants consume one 2g sachet containing 10e11 colony-forming units Bifidobacterium longum 1714 strain with maltodextrin and magnesium stearate on a daily basis over 1 year.
  Interventions: Dietary Supplement: Bifidobacterium longum 1714
- Placebo (Experimental): Participants consume one 2g placebo sachet containing maltodextrin and magnesium stearate.
  Interventions: Dietary Supplement: placebo sachet containing maltodextrin and magnesium stearate.

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum 1714 — This is a double-blind randomized placebo-controlled pilot study. Participants under extreme conditions of hypoxia, confinement and isolation receive Bifidobacterium longum 1714 on a daily basis over one year in order to test improvements on stress resilience and immune functions.
  Arms: Bifidobacterium longum 1714
Dietary Supplement: placebo sachet containing maltodextrin and magnesium stearate. — placebo sachet containing maltodextrin and magnesium stearate.
  Arms: Placebo

SUMMARY:
There is evidence to indicate that the gut microbiota has an effect on mental well-being and stress behaviours. This is highly relevant to both life on earth and spaceflight missions, in which mental well-being is crucial to mission success. Bifidobacterium longum 1714 (BL 1714), will be tested in the project ICELAND-2 in a double-blind, randomized placebo-controlled pilot study in crew members of the Antarctica station CONCORDIA in order to test stress resilience and possible outcomes on the immune system since the metabolic stress response and the immune system are closely interrelated. Crew members of CONCORDIA station have a prolonged stay (roughly 12 months) in a confined (antigen exposure restricted, overclean) and isolated environment, mimicking the situation of long-term space travel. ICELAND-2 will be conducted over three consecutive winter-over periods (3 years).

The project ICELAND-2:

1. evaluates the effect of the probiotic BL1714 on well-being regarding mood, social integration and stress and other parameters .
2. determines the effect of an antigen-limited environment like Concordia on gut microbiota, immune system and epigenetics.
3. examines the interaction between the factors mentioned in 1.
4. examines the role of nutrition intake and behaviour in the interplay mentioned above.

DETAILED DESCRIPTION:
EXPERIMENT CONCEPT

This is a double-bind, controlled pilot study where volunteers will receive a novel nutritional supplement powder (sachet, containing 1011 CFU Bifidobacterium longum 1714 (Alimentary 11 Health, Cork, Ireland) or placebo) once every day, to be taken in the morning with breakfastthroughout the year. The intervention starts for every participant at arrival (individual start). Using this study design, benefits of the probiotic on height adaptation can be also studied.

The experimental concept is based on the collection of biosamples (saliva, blood, stool) and some paper-pencil and documentary data only. Thereby, the interference of the project with the daily activities of the CONCORDIA crew is minimal. Both, female and male participants are included.

1. One blood, one saliva and one stool sample prior to the CONCORDIA stay, in addition to paper-pencil data collection once at the same time (-2 to 3 months prior to the stay - T Zero, BDC)
2. Three blood as well as a saliva samples (month 1, months 4 and 9, corresponding to T0, T4 and T9) during the CONCORDIA stay, as well as monthly collection of stool samples (months 1 to 9, T1 to T9), plus questionnaire data (paper-pencil data and/or online).
3. One blood, one saliva and one stool sample after the CONCORDIA stay, in addition to paper-pencil data collection once at the same time (3 to 6 months after the stay - T12)

Saliva Sampling: a standard saliva sampling kit (Oragene-DNA - OG-500, DNA Genotec, Ottawa, ON, Canada) will be used (see Figure 2).

Stool Sampling: a standard stool sampling kit (Sarstedt) will be used (see Figure 3) to retrieve 3 small samples from each stool, and stored in separated containers.

Feces Catcher: Paper-based stool collection aid (with instruction imprinted in variable language (FecesCatcher®) (Figure 4)

Blood sampling: Blood collection will be performed in two 5 ml heparinized tubes (total 10 ml for cell collection) and one dried tube of 5 ml per blood sampling. An adequate number of separation tubes and cryotubes for processing of blood will also be provided.

PROCEDURE OUTLINE

Saliva sampling: can be done at any time prior to the CONCORDIA stay, easiest during the pre-departure crew meeting. Saliva sampling will be repeated at month 4 and 9 as well as post CONCORDIA stay. Saliva samples do not need any preprocessing and can be stored at room temperature for the remaining time.

During the pre-departure meeting, a 1-hour interview related to nutritional habits (including gastrointestinal symptoms like bowel movements) should be done. Paper-pencil tests (1 hour) will be collected as well. This will include the Food Frequency Questionnaire (FFQ), the gastrointestinal symptom rating scale (GSRS) and a structured questionnaire related to previous illnesses, drug intake and medical treatments. The FFQ and the GSRS will be assessed in Concordia at the same times as the blood sampling is performed.

Stool sampling and short well-being assessment: Sampling (three aliquots, pea-size, in separate containers) can be done at the discretion of each participating CONCORDIA crew member once every month, but preferentially at approximately same day of the months each time. No coordinated sampling between crew members is needed, but the day should be noted on the sampling kits/diary. This should be supervised and documented by the ESA MD. Along with the stool sampling the participants will be asked to rate on a visual analogue scale mood, stress and social integrity. Additionally, the ESA MD will provide the information for every participant. This measure is needed as outcome for the RCT.

Food records: The ESA MD is asked to take pictures of meals/food/food condition on a regular base if possible. Most importantly, the MD should take standardized photos of the meals (of the last three days prior to the and the days of the stool sampling. The camera and storage devices have been handed out to the MD in Aosta, Italy.

Alternatively and/or in addition the cook will record his cooking activities.

T - 3 days before stool sampling:

ESA MD takes photo (with a reference 2 euro coin) of breakfast meal, lunch meal and dinner meal

T - 2 days before stool sampling:

ESA MD takes photo (with a reference 2 euro coin) of breakfast meal, lunch meal and dinner meal

T - 1 days before stool sampling:

ESA MD takes photo (with a reference 2 euro coin) of breakfast meal, lunch meal and dinner meal

Days of stool sampling:

ESA MD takes photo (with a reference 2 euro coin) of breakfast meal, lunch meal and dinner meal

Pre-processing of stool samples is not needed, samples are stored away at -50°C.

Blood sampling: Blood withdrawal for immune testing must be performed by a single phlebotomy, and can be performed at the time of programmed health checks of the CONCORDIA staff. Blood collection must be performed in two 5 ml heparinized tubes (total 10 ml for cell collection), and one dried tube of 5 ml for serum.

Pre-processing of the Blood Sample (to be performed by the ESA investigator physician)

For cognate immune functions, live cells are needed and must be frozen and stored in preserving conditions so they can be resuscitated after that. This means rapid processing after collection (within 4-6 hours), fast freezing and in preserving medium (with DMSO) below -40°C.

Blood Cell storage: Vacutainer® CPT™ Cell Preparation tubes with Sodium Heparin are provided to simplify cell preparation (Figure 5, left). CPT™ tubes directly contain ficoll (density buffer) and a gel ready for centrifugation. The blood is collected on the top of the gel like usual vacutainer tubes. Centrifugation will separate red blood cells, granulocytes (going below the gel) from mononuclear cells and plasma staying on the top. Mononuclear cells need washing in Sterile Hanks buffer (provided) and the pellet re-suspended in freezing buffer (provided) and directly frozen at least below 40°C.

ELIGIBILITY:
Inclusion Criteria:

Crew members of the Concordia station in Antarctica

Exclusion Criteria:

Participants which are not crew members of the Concordia station in Antarctica

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Expert rating by medical doctor on well-being of participant | up to 12 months
  The medical doctors will rate the well-being of participants structured using 10 visual analogue scales monthly. The scales comprise the topics stress, stress coping, mood and physical health. This Rating is done ahead of the participant ratings (see sec. outcomes)

SECONDARY OUTCOMES:
Participant rating on well-being | measurement monthly over 12 months
  The participants will perform a self-rating of their well-being using the same visual analogue scales as the medical doctor for the primary outcome.
Discrepancy between ratings on well-being | measurement monthly over 12 months
  The discrepancy between the expert-rating and the self-rating will be calculated
Gastrointestinal symptoms | Measurements at 1 day predeparture, in Antarctica at months 4,9 and 12 and 6 months postdeparture
  Gastrointestinal symptoms will be assessed using the gastrointestinal symptom rating scale
Gastrointestinal microbiota | stool samples collected at 1 day predeparture, in Antarctica monthly over 1 year and 6 months postdeparture
  Gastrointestinal microbiota composition and diversity measures analysed from stool samples using 16S rRNA sequencing and shotgun sequencing
Immune system | Measurements at 1 day predeparture, in Antarctica at months 4,9 and 12 and 6 months postdeparture
  Cognate immune system analyzed from blood samples using FACS
Epigenetics | Measurements at 1 day predeparture, in Antarctica at months 4,9 and 12 and 6 months postdeparture
  Histone modification and DNA methylation with focus on immune biology (DNA from saliva samples) using state of the art techniques e.g. Chromatin immunoprecipitation (ChIP)-based methods and high-performance liquid chromatography (HPLC), bisulfite sequencing, and CpG island microarrays.
Interaction between microbiota and immune biology (including epigenetics) | Measurements at 1 day predeparture, in Antarctica at months 4,9 and 12 and 6 months postdeparture
  Interaction between microbiota and immune biology (including epigenetics) by using novel bioinformatic and statistic models e.g. distance based redundancy analysis
Nutrition | FFQ: Measurements at 1 day predeparture, in Antarctica at months 4,9 and 12 and 6 months postdeparture
  Influence of nutrition and nutritional habits on healths using Food Frequency Questionnaires (FFQ) and standardized photographies of meals
Medical and psychological data records assessed by the medical doctors of the European Space Agency | 1 day Predeparture, Antarctica winterover of 12 months
  Medical and psychological data records assessed by the medical doctors of the European Space Agency
POMS | 1 day Predeparture, Antarctica winterover of 12 months
  Profile of mood states (POMS) questionnaire
PANAS | 1 day Predeparture, Antarctica winterover of 12 months
  Positive & negative affect schedule

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia Station, Concordia, Antarctica